CLINICAL TRIAL: NCT06220734
Title: Early Detection of the Effect of Irrigation Fluid on Extravascular Lung Water in Patients Undergoing Transurethral Resection of a Prostate Using Bedside Lung Ultrasound
Brief Title: Detection of the Effect of Irrigation Fluid on Extravascular Lung Water in Patients Undergoing TRUP Using Bedside Lung Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Monica Nabil Helmy Elcellini, Resident Doctor, Assiut University
Other Study IDs: US in Anesthesia
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: TUR Syndrome; Anesthesia
MeSH Terms: interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — None Retained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: transurethral resection of the prostate — transurethral resection of the prostate for indicated patients then US was done for early detection of fluid accumulation in the lungs

SUMMARY:
Early detection of fluid accumulation in alveolar, interstitial, and intracellular compartments of the lung due to intravascular absorption of irrigation fluid of TURP guided by lung ultrasound by detection of sonographic B lines.

DETAILED DESCRIPTION:
Endoscopic syndrome or TURP (transurethral resection of a prostate syndrome (TURP)) syndrome is an undesirable effect of prostatectomy through the urethra. The reason is that the lavage used in endoscopy is hypotonic fluid, without electrolytes absorbed into the lumen through the prostate venous sinuses, changing the circulating volume, disturbing the water balance of electrolytes, especially hyponatremia, and reducing serum osmolality, affecting on the cardiovascular system, respiratory and nervous system.1 Symptoms of TURP are often irregular, asynchronous, and nonspecific. Sometimes life-threatening complications such as sudden coma, heart failure, cardiovascular collapse and, respiratory failure2,3 are reported. Recent studies show that the incidence of TURP ranges from 0.78% to 1.4%. Although there are not many severe cases of TURP, the mortality rate is up to 25%.4,5

The TURP syndrome is a clinical diagnosis based upon a constellation of symptoms and signs associated with excessive absorption of irrigating fluid into the circulation. It comprises acute changes in intravascular volume, plasma solute concentrations, and osmolality, and direct effects of the irrigation fluid used (glycine and its metabolites in the UK, as glycine 1.5% is the most common irrigation fluid used). The effects are proportional to the volume of irrigating solution absorbed. The presentation is not always uniform, and milder cases may be unrecognized. Other types of endoscopic surgery that require the use of irrigation solution, e.g., hysteroscopy, may also give increase to the TURP syndrome.3

Mild-to-moderate TURP syndrome may occur in 1-8% of patients.3 The overall mortality is 0.2-0.8%. It may present as early as 15 min after resection starts or as late as 24 h after operation.6 Severe TURP syndrome is now rare; however, it carries a mortality of up to 25%.3

Irrigation fluid is absorbed at a rate of between 10- and 30-ml min-1 of operating time.6 Five to 20% of patients will absorb >1 litre.3

A higher rate of absorption is produced by several factors.

1. The pressure of the irrigation fluid. The height of the bag should be kept as low as possible to achieve adequate flow of fluid. Seventy centimeters are usually satisfactory. However, the surgeon will frequently stop and drain the bladder to remove chippings; during this time, the hydrostatic pressure within the bladder is low.
2. Low venous pressure, e.g., if the patient is hypovolemic or hypotensive.
3. Prolonged surgery, especially >1 h, although this is now uncommon.
4. Large blood loss, implying many open veins.
5. Capsular perforation, or bladder perforation, allowing a large volume of irrigation fluid into the peritoneal cavity, where it is rapidly absorbed.

Acute volume changes affect the cardiovascular system. The rapid absorption of a large volume of irrigation fluid can cause hypertension with reflex bradycardia and can precipitate acute cardiac failure and pulmonary oedema. The magnitude of the hypertension is not related to the volume of fluid absorbed.

Rapid equilibration of hypotonic fluid with the extracellular fluid compartment may precipitate sudden hypotension in association with hypovolemia. Hypotension and hypovolemia may be compounded by the sympathetic block of spinal anesthesia. This secondary phase at the end of the operation is often the first sign suggestive of the TURP syndrome.

The guidelines for intraoperative intravenous (IV) fluid administration are poorly defined, and fluid administration varies from restrictive to liberal fluid administration.[7] The goals of intraoperative fluid administration should be to maintain proper volume in the circulation to maintain adequate tissue perfusion. Traditionally, a large volume of fluid is infused intraoperatively[8] with the belief that overnight fasting and the effect of anesthesia on ongoing blood loss during surgery lead to hypovolemia that results in reduced circulatory volume and diminished tissue perfusion.[9,10] In contrast, inadequate fluid administration may lead to circulatory instability, compromised tissue perfusion and complications such as prerenal acute renal failure.[10-12] Liberal fluid administration has concerns about pulmonary congestion or oedema, decreased wound healing, decreased tissue oxygenation and delayed recovery.[7]

Over the past decade, ultrasound and particularly lung ultrasound (LUS) has rapidly gained increasing importance as a monitoring and diagnostic tool in the intensive care unit (ICU) (13)

Yet, for several lung disorders typically associated with intensive care settings such as pulmonary edema, pneumonia, or pleural effusions, LUS has recently proven its superiority over other diagnostic invasive and non-invasive imaging techniques such as chest radiography or physical examinations like auscultation. Specifically, LUS provides a higher diagnostic value, is more cost-effective and especially easy to perform directly at the patient's bedside (14-18).

Sonographic visualization of B-lines-originally termed as comet-tail artifacts arising vertically from the hyperechoic pleural line-represents a promising alternative for assessment of lung water.20 Scoring of B-lines is typically performed by their summation from different intercostal spaces.19 Most commonly recommended, an extensive 28-sector protocol of the antero-lateral chest is used for evaluation of quantitative B-lines score.21,22.

ELIGIBILITY:
Inclusion Criteria:

* • ASA Class I, II or III adult patients of age group 18-65 years.

  * Patient undergoing TURP.

Exclusion Criteria:

* • Patients unable to provide written consent.

  * Patients less than 18 years or above 65 years.
  * ASA Class IV.
  * Patients previously diagnosed to suffer from interstitial lung disease.
  * patients who will receive intraoperative diuretics

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men attended at assuit university hospital, for underwent transurethral resection of the prostate and fulfilled inclusion criteria
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-05 (Estimated); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative lung congestion quantified by number of sonographic B-lines in anterolateral lung ultrasound scan in patients undergoing TURP | 1 year
  Early detection of fluid accumulation in alveolar, interstitial, and intracellular compartments of the lung due to intravascular absorption of irrigation fluid of TURP guided by lung ultrasound by detection of sonographic B lines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gravenstein D. Transurethral resection of the prostate (TURP) syndrome: a review of the pathophysiology and management. Anesth Analg. 1997 Feb;84(2):438-46. doi: 10.1097/00000539-199702000-00037. No abstract available. PMID 9024044
- [Background] Gupta K, Rastogi B, Jain M, Gupta PK, Sharma D. Electrolyte changes: An indirect method to assess irrigation fluid absorption complications during transurethral resection of prostate: A prospective study. Saudi J Anaesth. 2010 Sep;4(3):142-6. doi: 10.4103/1658-354X.71505. PMID 21189849